CLINICAL TRIAL: NCT05194761
Title: Normal Saline Nebulization in Prevention of Extubation Failure in Neonates
Brief Title: Normal Saline Nebulization on Prevention of Extubation Failure in Neonates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Olivia Zakaria ,MSC, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AinShamsUPed
Record Dates: First submitted 2021-12-31; First posted 2022-01-18 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2021-11

CONDITIONS: Neonatal Respiratory Failure
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- using nebulization (Active Comparator): extubated neonates will be divided in two group , one will receive saline nebulization for 3 days postextubation ,
  Interventions: Drug: Normal saline
- No nebulization (No Intervention): the other group will only receive the standard only

INTERVENTIONS:
Drug: Normal saline — Using normal saline nebulization in neonates postextubation
  Arms: using nebulization

SUMMARY:
this study is about evaluating the effect of using normal saline nebulization in preventing re-intubation in extubated neonates , provided that the cause of intubation is mainly due to respiratory cause

DETAILED DESCRIPTION:
Using nebulization is of great debate in neonates especially post extubation as neonates have physiological characteristics such as difficult airway maintenance and clearance, smaller airway caliber, compliant chest wall, poor airway stability, and lower functional residual capacity that account for the diminished delivery of inhaled aerosol.

Nebulized normal saline has historically been used as a placebo typically in studies examining bronchodilator medications and sputum expectorants or used as a carrier to medications. Nowadays, normal saline is a method of enhancing mucociliary clearance has become a clinically accepted adjunct to physiotherapy in the treatment of many chronic lung conditions .

the effect of whether or not nebulization really improves the lung condition is evaluated by lung ultrasound ,It is not only useful in predicting failure of non-invasive ventilation and the need for invasive ventilation, but also has a great value in anticipating extubation success In general, patients with lower lung ultrasound scores show a better chance of extubation success. Each lung will be divided into 3 areas (upper anterior, lower anterior, and lateral) and will be examined using a linear microprobe through both transverse and longitudinal scans. For each lung area, a 0- to 3-point score was given (total score ranging from 0-18).

ELIGIBILITY:
Inclusion Criteria:

* Ventilated babies with primary respiratory disease as the provisional and primary cause of intubation immediately post-extubation.

Exclusion Criteria:

* Neurological, cardiac, surgical or metabolic problems affecting their respiration.

Upper obstructive air way disease that might affect the success of extubation.

Max Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-10-03 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Reintubation by 72 hours post-extubation | within 72 hours
  Number of participants with successful extubation

SECONDARY OUTCOMES:
Lung ultrasound score | 72 hours
  Number of participants with higher score may have worse prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Rania ElFarrash, Prof., Study Chair — Ain Shams University; Ibrahim Abuseif, Prof., Study Chair — Ain Shams University
Locations (1):
- AinShams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided